CLINICAL TRIAL: NCT04695080
Title: ChariotMS - A National (UK) Phase IIb, Multi-centre, Randomised, Double-blind, Placebo Controlled (1:1) Efficacy Trial With Cost-utility Analysis of Cladribine Tablets (3.5mg/kg Over Two Years) in People With Advanced Multiple Sclerosis. Is Cladribine Superior to Placebo in Protecting Upper Limb Function?
Brief Title: ChariotMS - Cladribine to Halt Deterioration in People With Advanced Multiple Sclerosis
Acronym: ChariotMS
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Merck Serono Limited, UK (Industry); Multiple Sclerosis Society of Great Britain & Northern Ireland (Unknown); National Multiple Sclerosis Society (Other); Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 258909; 2018-005038-39 (EudraCT Number)
Record Dates: First submitted 2020-11-06; First posted 2021-01-05 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Advanced Multiple Sclerosis; Progressive Multiple Sclerosis
Keywords: Multiple Sclerosis; Progressive multiple sclerosis; Advanced multiple sclerosis; Upper limb function; Cladribine; Quality of life; Cognition; Health Economics; Biomarkers; Neurofilament light chain; B cells; Lymphocytes; Magnetic Resonance Imaging (MRI)
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis; Charcot-Marie-Tooth disease, Type 1F | interventions — Cladribine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cladribine (MAVENCLAD®) (Active Comparator)
  Interventions: Drug: Cladribine (MAVENCLAD®)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cladribine (MAVENCLAD®) — Cladribine (MAVENCLAD®) 3.5mg/kg, administered as weight-adjusted 10mg tablets in two treatment courses (12 months apart) lasting 8- 10 days each.
  Cladribine (MAVENCLAD®) 10mg available in blister packs of 1 tablet, 4 tablets and 6 tablets.
  Arms: Cladribine (MAVENCLAD®)
Drug: Placebo — Placebo administered as weight adjusted tablets in two treatment courses (12 months apart) lasting 8-10 days each.
  Placebo 10mg available in blister packs of 1 tablet, 4 tablets and 6 tablets.
  Arms: Placebo

SUMMARY:
MS is a chronic inflammatory and degenerative disease of the central nervous system (CNS) affecting more than 120,000 people in the UK.and 2.5 million people worldwide.

Without disease modifying treatment (DMT),the majority of people with MS (pwMS) will develop significant disability within 10 years of onset, and 50% will require wheelchair assistance within 20 years. convenient, highly effective and CNS penetrant DMT for patients with relapsing multiple sclerosis (pwRMS) administered in short (8-10 days/year over 2 years) treatment courses.

It effectively depletes B cells, particularly Memory B cells, a likely key mechanism of disease control in MS. Cladribine is the investigational product in this study as it not currently used to treat patients with an EDSS of 6.5 - 8.5. This is a multi-centre, randomised double-blind placebo-controlled phase IIb to test cladribine tablets (MAVENCLAD®) (3.5mg/kg over 24 months) for safety, efficacy, and cost effectiveness, and to advance mechanistic understanding of its action in people with advanced MS (pwAMS).

ELIGIBILITY:
Inclusion criteria:

1. pwAMS aged 18+ years with an EDSS of 6.5-8.5 (inclusive)
2. History of bowel cancer screening for men, and women and cervical and breast cancer screening for women as per NHS recommended guidelines https://www.nhs.uk/conditions/nhs-screening/.
3. Ability to complete the 9HPT with at least one upper limb within 180 seconds. The average score of both attempts for each hand should be used to assess eligibility.
4. Confirmation of MS diagnosis according to the McDonald Criteria (2017) Thompson et al. 2018).
5. In the judgement of the investigator, evidence of deterioration of upper limb function during the 2 years running up to the screening date.

Exclusion Criteria

1. Participants with known hypersensitivity to Cladribine of any grade (as per CTCAE grading system) should be excluded
2. Any uncontrolled diabetes, arterial hypertension and hypercholesterolaemia as determined by PI or delegated sub-investigator
3. A history of stroke and/or myocardial infarction
4. Moderate to severe renal impairment (creatinine clearance <60 ml/min)
5. Moderate to severe hepatic impairment (Child-Pugh score >6)
6. Significant comorbidity, e.g. cardiac failure, renal failure, malignancy, or other health condition that in the view of the PI or delegated sub-investigator precludes participation. Patients who, following discussion with their cancer treatment team, are deemed to be cured from malignancy, may be eligible to participate as per the clinical judgement of the local PI.
7. Pregnancy including planning to father a child or breastfeeding
8. Body weight less <40kg
9. Unwillingness to use effective contraception throughout the trial period until at least six months after the last administration of IMP. This is not applicable for post-menopausal women
10. Acute infection (uncontrolled)
11. Infection with Human Immunodeficiency Virus 1 and/or 2
12. Active chronic infection (Syphilis, Tuberculosis, Hepatitis). Patients with active TB will be excluded. However, patients who have a positive IGRA, Elispot or Quantiferon test, but exhibit no symptoms for TB and evidence of a normal Chest X Ray, can be included in the study as per judgement of the local PI and after clarification with the CI.
13. Precancerous condition
14. Total lymphocyte count <1.0*109/L
15. Seronegativity for varicella zoster virus. Potential participants who are IgG negative may undergo vaccination, and can be screened again once full course has been completed.

    Seronegativity for all of the following: measles, mumps, rubella. Potential participants who are IgG negative for all 3 viruses, may undergo vaccination and can be screened again once full course has been completed.
16. Relapse within six months before screening
17. Inability to complete an MRI (contraindications for MRI, including but not limited to, MRI-non-compatible pacemaker, cochlear implants, intracranial vascular clips, surgery within 6 weeks of entry in the study, coronary stent implanted within 8 weeks prior to the time of the intended MRI, severe anxiety or claustrophobia etc.) or contraindication to Gd administration.
18. Treatment with steroids due to MS relapse/progression within three months of screening. pwAMS who fall in this category may undergo a further screening visit once the three months' window has expired and may be included if no steroid treatment has been administered in the intervening period. If for any reason a participant is unable to have a baseline MRI scan (due for safety reasons), this MRI scan may be omitted and a recent 'historical' MRI scan (collected within the 3 months preceding the first IMP dose dispensing at Baseline visit) can be used at the CI's discretion. This will need to be assessed by the CI case by case basis. The review of the historical MRI scan to exclude PML should be clearly documented in the subject's electronic health records prior to the first IMP dose dispensing at Baseline visit.
19. Treatment with any interferon-beta, glatiramer acetate, teriflunomide, leflunomide or dimethyl-fumarate within three months before screening.
20. Treatment with natalizumab, fingolimod, siponimod, ponesimod, ozanimod (or other Sphingosine-1-phosphate receptor modulators) within three months of screening.
21. Treatment with azathioprine, methotrexate, or cyclosporine within six months before screening.
22. pwAMS treated with teriflunomide will need to undergo accelerated elimination of the compound before being considered (Research and Case Medical Research 2019).
23. Treatment with haematopoietic stem cell transplantation (HSCT), mitoxantrone, cyclophosphamide, cladribine, alemtuzumab, or another B cell depleting compound, such as rituximab, ocrelizumab, ublitiuximab, ofatumumab, or biosimilars, unless the participant concerned has a memory B cell level of ≥20% of the CD19+ population in the peripheral blood. Such a level would normally not be expected earlier than a minimum of six months after the last drug administration. Participants who underwent such treatment will therefore have to be tested for their CD19+/CD27+ memory B cell level at screening.
24. Treatment with fampridine: If they are already on treatment for at least one month, participants should continue throughout the trial. However, starting continuous fampridine treatment after signing the consent sheet will lead to exclusion from treatment with IMP/placebo.
25. Concurrent participation or previous participation within the last 6 months in another clinical trial of an IMP or medical device.
26. Unable to swallow tablets

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The 9-HPT peg speed (tasks/second) at 24 months | 24 months
  To establish whether there is efficacy superiority of cladribine tablets over placebo in reducing deterioration of upper limb function in pwAMS.
  To investigate whether cladribine tablets 3.5mg/kg over 24 months is an effective DMT in pwAMS as measured using the 9-hole peg test (9HPT) peg speed at 24 months.
9-HPT proportion of patients who do not deteriorate at 24 months | 24 months

SECONDARY OUTCOMES:
Change over 24 months of the study in clinical outcome measure: EDSS | Screening, Month 6, 12, 18 and 24
  The proportion of the cladribine versus placebo arms with an increase of >=0.5 in EDSS score over 24 months.
Change over 24 months of the study in clinical outcome measure: ARAT | Screening, Month 6, 12, 18 and 24
  ARAT (Upper Limb Function Test) upper limb function test score
Change over 24 months of the study in clinical outcome measure: ABILHAND | Screening, Month 6, 12, 18 and 24
  ABILHAND score for manual ability
Change over 24 months of the study in clinical outcome measure: T25ftWT | Screening, Month 6, 12, 18 and 24
  Lower Limb Function: The T25ftWT (Timed 25 foot walk test) will be collected in all pwAMS able to walk the required distance twice.
Change over 24 months of the study in clinical outcome measure: SLCVA | Screening, Month 6, 12, 18 and 24
  SLCVA (Sloan low contrast letter visual acuity) score.
Change over 24 months of the study in clinical outcome measure: MSIS-29v2 | Screening, , Month 6, 12, 18 and 24
  MSIS-29v2 (Multiple Sclerosis Impact Scale) quality of life score
Change over 24 months of the study in clinical outcome measure: SDMT | Screening, Month 6, 12, 18 and 24
  SDMT (The Symbol Digit Modalities Test) score.
Change over 24 months of the study in clinical outcome measure: NFI-MS | Screening, Month 6, 12, 18 and 24
  NFI-MS (Neurological Fatigue Index-Multiple Sclerosis) score.
Change over 24 months of the study in clinical outcome measure: EuroQoL EQ-5D-5L | Screening, Month 6, 12, 18 and 24
  Cost-utility: Patient's generic health-related quality of life, measured using the EuroQoL EQ-5D-5L and, separately, carer's generic health-related quality of life, measured using the EuroQoL EQ-5D-5L, health and social care and other costs.
Change over 24 months of the study in clinical outcome measure: EuroQoL EQ-5D-5L | Screening, Month 6, 12, 18 and 24
  Cost-utility: Carer's generic health-related quality of life, measured using the EuroQoL EQ-5D-5L
Change over 24 months of the study in clinical outcome measure: EuroQoL EQ-5D-5L | Screening, Month 6, 12, 18 and 24
  Cost-utility: health and social care and other costs.
Change over 24 months of the study in clinical outcome measure: WPAI-GH | Baseline, Month 6, 12, 18 and 24
  WPAI-GH (Work Productivity and Activity Impairment Questionnaire: General Health V2.0 (WPAI:GH) score
Safety/occurrence of adverse events | Through study completion, an average of 24 months
  Safety:
  * Any AEs/SAEs,
  * Lymphopenia (peripheral blood lymphocyte counts),
  * Severe infections,
  * Malignancies.
  * Pregnancies
  * Special situations (e.g. overdose)
Preventing loss of brain volume | Screening, Month 6 and 24
  (MRI) Change over 24 months of the study in ventricular volume assessed using the VIENA technique.
Preventing loss of brain volume | Screening, Month 6 and 24
  (MRI) Change over 24 months in brain volume assessed using the "Structural Image Evaluation, using Normalisation, of Atrophy" (SIENA) technique
Preventing loss of spinal cord cross sectional area | Screening, Month 6 and 24
  (MRI) Change in the total cross-sectional area of spinal cord (at level C2) over 24 months
Preventing new focal demyelinating lesions and T2 burden of disease increase. | Screening, Month 6 and 24
  (MRI) Total number of new focal demyelinating brain lesions over 24 months
Preventing new hypo-intense lesions ("black holes") on T1 weighted MRI | Screening, Month 6 and 24
  (MRI) Total number of new hypo-intense T1 lesions over 24 months
Degree of unblinding | Month 24
  To determine the perception of treatment allocation for both participants and trial teams at 24 months.

OTHER OUTCOMES:
To determine if cladribine correlates with memory Bcell count. | Screening, Month 12 and 24
  Memory B-Cell (total number and percentage of CD19+ cell count) and its association with upper limb function as measured using 9HPT speed.
To determine association between Memory B cell count and 9HPT speed. | Screening, Month 6, 12, 18 and 24
  9HPT speed
To determine association between Memory B cell count and 9HPT speed. | Screening, Month 6, 12, 18 and 24
  ARAT score
To determine association between Memory B cell count, upper limb function and s-NfL level. | Screening, Month 12 and 24
  Serum-NfL at 6 and 24 months compared to baseline.
To determine effects of IMP on cortical and deep grey matter volumes, thalamic, hippocampal and ventricular volumes (VIENA) and slowly expanding (i.e. chronically active) lesions. | Screening, Month 6 and 24
  (MRI) Change over 24 months of the study in cortical brain volume
To determine effects of IMP on cortical and deep grey matter volumes, thalamic, hippocampal and ventricular volumes (VIENA) and slowly expanding (i.e. chronically active) lesions. | Screening, Month 6 and 24
  (MRI) Change over 24 months of the study in thalamic brain volume
To determine effects of IMP on cortical and deep grey matter volumes, thalamic, hippocampal and ventricular volumes (VIENA) and slowly expanding (i.e. chronically active) lesions. | Screening, Month 6 and 24
  (MRI) Change over 24 months of the study in hippocampal brain volume
To determine effects of IMP on cortical and deep grey matter volumes, thalamic, hippocampal and ventricular volumes (VIENA) and slowly expanding (i.e. chronically active) lesions. | Screening, Month 6 and 24
  (MRI) Change over 24 months of the study in new slowly expanding/evolving lesions (SELs)

CONTACTS AND LOCATIONS:
Locations (22):
- United Kingdom (22):
  - Queens University Belfast (Belfast Health and Social Care Trust), Belfast
  - University Hospitals Birmingham NHS Foundation Trust, Queen Elizabeth Hospital Birmingham, Birmingham
  - Cardiff University Hospital, Cardiff
  - University Hospitals of Coventry and Warwickshire NHS Trust, Coventry
  - Anne Rowling Clinic, University of Edinburgh, Edinburgh
  - Queen Elizabeth University Hospital Glasgow, Glasgow
  - University Hospital Hairmyres, NHS Lanarkshire, Glasgow
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Walton Centre NHS Trust, Liverpool
  - Royal London Hospital, London
  - Royal Free London NHS Foundation Trust, London
  - Queen's Hospital (Havering and Redbridge University Hospitals NHS Trust), London
  - Lewisham and Greenwich NHS Trust, London
  - St George's University Hospitals NHS Foundation Trust, London
  - Luton and Dunstable Hospital, Luton
  - Salford Royal Hospital NHS Trust, Manchester
  - Aneurin Bevan University Health Board, Newport
  - Nottingham University Hospital (Nottingham University Hospitals NHS Trust), Nottingham
  - University Hospitals Plymouth NHS Trust, Plymouth
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - University Hospitals of North Midlands NHS Trust, Stoke-on-Trent
  - Morriston Hospital, Swansea, Swansea

IPD SHARING:
Plan to Share IPD: No